CLINICAL TRIAL: NCT06130319
Title: Correlation of Disease Management and Quality of Life in Patients With Chronic Heart Failure and Their Family Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1051-01
Record Dates: First submitted 2023-11-02; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to investigate the current status of disease management and quality of life of patients with chronic heart failure and their family caregivers, explore the relationship between the two sides of disease management and quality of life, help nurses identify the influencing factors of quality of life of patients with chronic heart failure and their family caregivers, and carry out family-centered care in the future. This study intends to investigate the current status of disease management and quality of life of patients with chronic heart failure and their family caregivers, explore the relationship between disease management and quality of life of both sides, and help nurses identify the influencing factors affecting the quality of life of patients with chronic heart failure and their family caregivers, so as to carry out family-centered care in the future. To provide theoretical basis for improving the quality of life of both parties.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of Chinese Guidelines for the diagnosis and treatment of heart failure
2. the duration of chronic heart failure was ≥3 months;
3. have certain reading, comprehension and expression ability, and can complete the questionnaire independently or with the guidance of the researcher;
4. Informed and agreed to participate in the investigation

Exclusion Criteria:

* In the acute stage of the disease, such as acute heart failure attack or complicated with severe pulmonary infection, liver and kidney function damage, etc.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients in the department of cardiology of a tertiary hospital in Guangzhou
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
the quality of life questionnaire | 10 months
  Quality of life refers to the subjective feelings of individuals about their own goals, expectations, standards, and life situations related to the things they care about in different cultures and value systems

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, China